CLINICAL TRIAL: NCT02671851
Title: Ultrasound-Guided Bilateral Thoracic Paravertebral Blocks as an Adjunct to General Anaesthesia in Patients Undergoing Reduction Mammoplasty: A Historical Cohort Study
Brief Title: Ultrasound-Guided Thoracic Paravertebral Blocks in Patients Undergoing Reduction Mammoplasty
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emine Aysu Salviz, MD, M.D., Attending Anesthesiologist, Istanbul University
Other Study IDs: 2016/83
Record Dates: First submitted 2016-01-22; First posted 2016-02-02 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Pain, Postoperative
Keywords: Thoracic Paravertebral Blocks; Ultrasound Guidance; Reduction Mammoplasty; Time to First Pain; Postoperative Analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dipyrone; Acetaminophen; Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thoracic paravertebral blocks (TPVBs): Patients received bilateral single injection ultrasound-guided TPVBs at the level of T3-T4 with 20 mL bupivacaine 0.375% as an adjunct to general anaesthesia. IV metamizole sodium and paracetamol were rescue analgesics.
  Interventions: Drug: Thoracic paravertebral blocks (TPVBs)
- IV metamizole sodium, paracetamol: Patients received only standardized general anaesthesia. IV metamizole sodium and paracetamol were rescue analgesics.
  Interventions: Drug: IV metamizole sodium, paracetamol

INTERVENTIONS:
Drug: Thoracic paravertebral blocks (TPVBs) — Patients received bilateral single injection ultrasound-guided TPVBs with 20mL bupivacaine 0.375% at the level of T3-T4 as an adjunct to GA, intraoperative fentanyl and postoperative tramadol, metamizole sodium and paracetamol were used.
  Other Names: Bupivacaine,fentanyl,tramadol,metamizole sodium,paracetamol
  Groups: Thoracic paravertebral blocks (TPVBs)
Drug: IV metamizole sodium, paracetamol — Patients received only standardized GA, intraoperative fentanyl and postoperative tramadol, metamizole sodium and paracetamol were used.
  Other Names: Fentanyl,tramadol,metamizole sodium,paracetamol
  Groups: IV metamizole sodium, paracetamol

SUMMARY:
Background: Thoracic paravertebral blocks (TPVBs) have been effective for postoperative analgesia in mastectomy, thoracic and video-assisted thoracic surgeries.

Objective: To assess whether addition of ultrasound-guided TPVBs to general anaesthesia (GA) could postpone time to first pain and improve postoperative analgesia in patients undergoing bilateral reduction mammoplasty.

Design: A historical cohort study. Patients: Of the 70 female patients who underwent bilateral reduction mammoplasty, 64 patients had complete data in the acute pain/regional anaesthesia database.

Intervention: Thirty patients, received only GA, were included in Group GA. Thirty-four patients, received bilateral single injection ultrasound-guided TPVBs with 20 mL bupivacaine 0.375% as an adjunct to GA, were included in Group TPVBs. Patients in both groups were administered intraoperative fentanyl if heart rate or mean arterial pressure increased >20% above pre-induction values, postoperative tramadol 1mg/kg in the postoperative care unit (PACU) if numeric rating scale (NRS) was ≥4, and rescue analgesics as metamizole sodium 4x1g and/or paracetamol 3x1g on wards (NRS≥4).

Main outcome measures: The primary endpoint was time to first pain after the surgery. Secondary endpoints were intra- and postoperative opioid and other rescue analgesic requirements, length of stay in the PACU, pain scores, incidence of postoperative nausea and vomiting (PONV), and patient and surgeon satisfaction through the postoperative first 2 days.

DETAILED DESCRIPTION:
Background: Thoracic paravertebral blocks (TPVBs) have been effective for postoperative analgesia in mastectomy, thoracic and video-assisted thoracic surgeries.

Objective: The objective was to assess whether addition of ultrasound-guided TPVBs to general anaesthesia (GA) could postpone time to first pain and improve postoperative analgesia in patients undergoing bilateral reduction mammoplasty.

Design: A historical cohort study. Patients: Of the 70 female patients who underwent bilateral reduction mammaplasty, 64 patients had complete data in the acute pain/regional anaesthesia database.

Intervention: Standard monitoring was applied before any anesthetic techniques were performed. All patients were given sedation in the form of midazolam 1-2 mg and fentanyl 50-100 µg. Patients underwent bilateral reduction mammaplasty were distributed to two groups due to their data: 1) Patients received only general anaesthesia (GA) were included in Group GA, and 2) Patients received preoperative US-guided TPVBs as an adjunct to GA were included in Group TPVBs. Thirty patients were in Group GA. Thirty-four patients who were in Group TPVBs received bilateral single injection ultrasound-guided TPVBs with 20 mL bupivacaine 0.375% (20 mL per injection) at the level of T3-4, as an adjunct to GA. Patients in both groups were administered intraoperative fentanyl if heart rate or mean arterial pressure increased >20% above pre-induction values. They also received postoperative tramadol 1mg/kg in the postoperative care unit (PACU) and rescue analgesics as metamizole sodium 4x1g and/or paracetamol 3x1g on wards, if numeric rating scale (NRS) was ≥4.

Main outcome measures: The primary endpoint was time to first pain after the surgery. Secondary endpoints were intra- and postoperative opioid and other rescue analgesic requirements, length of stay in the PACU, pain scores, incidence of postoperative nausea and vomiting (PONV), and patient and surgeon satisfaction through the postoperative first 2 days.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients who underwent bilateral reduction mammoplasty

Exclusion Criteria:

* Patients with deficient data

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients undergoing bilateral reduction mammoplasty
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Time to first pain | 0-48 hours
  Postoperative first pain description NRS ≥4

SECONDARY OUTCOMES:
Fentanyl use | During the surgery
  Intraoperative fentanyl was used if heart rate or mean arterial pressure increased >20% above preinduction values
Tramadol use | 0-2 hours
  Postoperative pain NRS ≥4 in the postoperative care unit
Rescue analgesic requirement | 0-48 hours
  Postoperative pain NRS ≥4 on the wards
Length of stay in the PACU | 0-2 hours
  White's Fast-Tracking Scoring System ≥12 was used for PACU discharge with no score of <1 in any category
Pain (NRS) scores | 0-48 hours
  Numeric rating scale (NRS) pain scores (0: no pain, 10: worst pain imaginable)
Incidence of Postoperative nausea and vomiting (PONV) | 0-48 hours
  Incidence of PONV
Patient satisfaction (Satisfaction scores) | 0-48 hours
  Satisfaction scores (0: very unsatisfied, 3: very satisfied)
Surgeon satisfaction (Satisfaction scores) | 0-48 hours
  Satisfaction scores (0: very unsatisfied, 3: very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Emine A Salviz, MD, Principal Investigator — Design and conduct the study, review and analyze the data, and write the manuscript
Locations (1):
- Istanbul University, Department of Anaesthesiology, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaya FN, Turker G, Mogol EB, Bayraktar S. Thoracic paravertebral block for video-assisted thoracoscopic surgery: single injection versus multiple injections. J Cardiothorac Vasc Anesth. 2012 Feb;26(1):90-4. doi: 10.1053/j.jvca.2011.09.008. Epub 2011 Nov 4. PMID 22055006
- [Result] Kaya FN, Turker G, Basagan-Mogol E, Goren S, Bayram S, Gebitekin C. Preoperative multiple-injection thoracic paravertebral blocks reduce postoperative pain and analgesic requirements after video-assisted thoracic surgery. J Cardiothorac Vasc Anesth. 2006 Oct;20(5):639-43. doi: 10.1053/j.jvca.2006.03.022. Epub 2006 Aug 8. PMID 17023279
- [Result] Moller JF, Nikolajsen L, Rodt SA, Ronning H, Carlsson PS. Thoracic paravertebral block for breast cancer surgery: a randomized double-blind study. Anesth Analg. 2007 Dec;105(6):1848-51, table of contents. doi: 10.1213/01.ane.0000286135.21333.fd. PMID 18042892
- [Result] Terheggen MA, Wille F, Borel Rinkes IH, Ionescu TI, Knape JT. Paravertebral blockade for minor breast surgery. Anesth Analg. 2002 Feb;94(2):355-9, table of contents. doi: 10.1097/00000539-200202000-00023. PMID 11812698
- [Result] Klein SM, Bergh A, Steele SM, Georgiade GS, Greengrass RA. Thoracic paravertebral block for breast surgery. Anesth Analg. 2000 Jun;90(6):1402-5. doi: 10.1097/00000539-200006000-00026. PMID 10825328